CLINICAL TRIAL: NCT07388160
Title: Evaluation of Preoperative and Postoperative Serum BDNF, IL-1β, and HMGB1 Levels and Cognitive Changes in Patients Undergoing General Anesthesia: Differences Between Patients With No Prior General Anesthesia and Those With Multiple Anesthesia Exposures
Brief Title: Neuroinflammatory Biomarkers After General Anesthesia: A Comparison Study
Status: Not yet recruiting | Type: Observational
Sponsor: University of Health Sciences Balikesir Hospital Eduation and Research (Other Government)
Collaborators: Malatya Turgut Ozal University (Other)
Responsible Party: Sponsor
Other Study IDs: s.kutlusoy
Record Dates: First submitted 2026-01-23; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Anesthesia; Neuroinflammation; Cognitive Disorders
Keywords: Brain Derived Neurotrophic Factor; Interleukin-1 beta; General Anesthesia; Neuroinflammation; Cognitive Dysfunction; Biomarkers; Sevofluran; Inflammatory Cytokines; Anesthesia Neurotoxicity
MeSH Terms: conditions — Neuroinflammatory Diseases; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- No Previous General Anesthesia: Healthy volunteers aged 18-65 years who have never undergone general anesthesia. This control group will undergo elective cholecystectomy surgery under general anesthesia. Blood samples will be collected preoperatively and 24 hours postoperatively to measure serum BDNF, IL-1β, and HMGB1 levels. Cognitive function will also be assessed at both time points.
- Previous General Anesthesia Exposure: Patients aged 18-65 years scheduled for elective cholecystectomy who have received general anesthesia at least once or multiple times in the past. Blood samples will be collected preoperatively and 24 hours postoperatively to measure serum BDNF, IL-1β, and HMGB1 levels. Cognitive function will also be assessed at both time points. This group will be compared with the control group to evaluate the impact of repeated anesthesia exposure on neuroinflammatory biomarkers and neurotrophic balance.

SUMMARY:
This prospective, observational study investigates the impact of repeated general anesthesia exposure on neuroinflammatory biomarkers and neurotrophic factors. The study will enroll 160 adult patients (aged 18-65 years) scheduled for elective cholecystectomy surgery, divided into two groups: patients with no previous general anesthesia exposure (n=80) and patients with at least one or more previous general anesthesia exposures (n=80).

Serum levels of Brain-Derived Neurotrophic Factor (BDNF), Interleukin-1 beta (IL-1β), and High Mobility Group Box 1 (HMGB1) will be measured using ELISA method at two time points: preoperatively (baseline) and 24 hours postoperatively. Cognitive function will also be assessed at both time points.

The primary objective is to evaluate whether multiple exposures to general anesthesia lead to significant differences in serum BDNF, IL-1β, and HMGB1 levels, reflecting changes in neurotrophic balance and neuroinflammatory response. This study aims to provide insights into the potential biochemical mechanisms underlying anesthesia-related cognitive changes and contribute original clinical data to the current literature on general anesthesia safety and neurobiological effects.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Scheduled for elective cholecystectomy surgery
* Either no previous general anesthesia exposure OR at least one or more previous general anesthesia exposures
* Ability to provide informed consent
* American Society of Anesthesiologists (ASA) physical status I-II

Exclusion Criteria:

* Chronic neurological diseases (Alzheimer's disease, Parkinson's disease, multiple sclerosis, etc.)
* Psychiatric illness requiring medication
* Metabolic syndrome (diabetes mellitus, hypertension, cardiac disease)
* Chronic inflammatory diseases (rheumatoid arthritis, systemic lupus erythematosus, etc.)
* Corticosteroid or immunosuppressive therapy within the last 6 months
* Patients requiring intensive care admission
* Pregnancy or breastfeeding
* Known allergy to anesthetic agents
* Inability to provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will enroll adult patients aged 18-65 years scheduled for elective cholecystectomy surgery at Malatya Turgut Özal University Training and Research Hospital. Participants will be divided into two groups based on their previous general anesthesia exposure history: (1) patients with no prior general anesthesia exposure (control group, n=80), and (2) patients with at least one or more previous general anesthesia exposures (study group, n=80). Healthy volunteers with no previous surgical or anesthesia history will comprise the control group, while patients with previous surgical procedures requiring general anesthesia will comprise the study group. Both groups will be matched for age and body mass index. Participants with chronic neurological diseases, psychiatric disorders, metabolic syndrome, chronic inflammatory conditions, or recent immunosuppressive therapy will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2026-01-25 (Estimated); Primary Completion 2026-08-25 (Estimated); Study Completion 2026-09-25 (Estimated)

PRIMARY OUTCOMES:
Change in Serum BDNF Levels | Preoperative (baseline) and 24 hours postoperative
  Change in serum Brain-Derived Neurotrophic Factor (BDNF) concentration measured by ELISA method, comparing preoperative baseline levels with postoperative levels at 24 hours
Change in Serum HMGB1 Levels | Preoperative (baseline) and 24 hours postoperative
  Change in serum High Mobility Group Box 1 (HMGB1) concentration measured by ELISA method, comparing preoperative baseline levels with postoperative levels at 24 hours
Change in Serum IL-1β Levels | Preoperative (baseline) and 24 hours postoperative
  Change in serum Interleukin-1 beta (IL-1β) concentration measured by ELISA method, comparing preoperative baseline levels with postoperative levels at 24 hours

SECONDARY OUTCOMES:
Correlation Between Biomarkers | At 24 hours postoperative
  Analysis of correlations between serum BDNF, IL-1β, and HMGB1 levels to evaluate the relationship between neurotrophic balance and systemic inflammatory response following general anesthesia
Comparison Between Single vs Multiple Anesthesia Exposure Groups | Preoperative (baseline) and 24 hours postoperative
  Statistical comparison of serum BDNF, IL-1β, and HMGB1 levels between patients with no previous general anesthesia exposure and those with previous general anesthesia exposure(s)

CONTACTS AND LOCATIONS:
Overall Officials: sevgi kutlusoy, Assoc. Prof. Dr., Study Chair — Saglik Bilimleri Universitesi

IPD SHARING:
Plan to Share IPD: Undecided
The decision to share individual participant data (IPD) will be made after consultation with the institutional ethics committee and upon completion of primary analyses. Any data sharing will be contingent upon appropriate ethical approval, participant consent provisions, and establishment of a formal data sharing agreement. The final decision will be determined based on ethical, legal, and privacy considerations specific to the Turkish healthcare system and institutional policies.